CLINICAL TRIAL: NCT04974918
Title: The Reliability and Versatility of Facial Artery Perforator-Based Nasolabial Flaps in The Reconstruction of Lip Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Ahmed, resident doctor at plastic surgery sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-07-07
Record Dates: First submitted 2021-07-16; First posted 2021-07-23 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Lip Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Facial Artery Perforator-Based Nasolabial Flaps in The Reconstruction of Lip defects (Experimental): participants will be chosen according to liable age and information will be given about complications
  Interventions: Procedure: Facial Artery Perforator-Based Nasolabial Flaps in The Reconstruction of large Lip defects post traumatic or post tumor resection.

INTERVENTIONS:
Procedure: Facial Artery Perforator-Based Nasolabial Flaps in The Reconstruction of large Lip defects post traumatic or post tumor resection. — A perforator near the defect was selected to accomplish a sufficient arc of rotation without tension. The flap was designed to cover the defect based on one perforator and to hide the donor site in the nasolabial fold. An incision on one side of the flap was made to the subcutaneous tissue. Undermining of the flap until the perforators were identified. After the perforators were identified, the flap was redesigned and an incision was made circumferentially. Dissection of the pedicle was performed until tension-free transposition was done to cover the defect, and the distal perforators were sacrificed to help flap movement.

SUMMARY:
Nasolabial flaps have limited mobility and may need two stages, mostly for intraoral defects .The facial artery perforator-based flap is the first true perforator flap in the face. It allows one-stage reconstruction and allows freedom in flap design.

The nasolabial perforator flap has certain advantages such as repair using a similar tissue, a wider rotation arc around the pedicle compared to the other regional flaps, and the primary closure of the donor area.

DETAILED DESCRIPTION:
Recently, perforator flaps have become popular in many areas of reconstructive surgery. They provide design freedom and reduce donor-site morbidity. Many traditional local flaps including nasolabial flaps are based on the use of the axial facial artery with multiple perforators. Flaps based on one perforator of the facial artery have been introduced and are used more frequently because of their advantages over perforator flaps.

According to recent literatures, facial artery provides numerous cutaneous perforators, on which skin flaps can be islanded, with greater mobility and liability for reconstruction of small-to-moderate-sized intraoral and facial defects in one stage. .

Multiple perforators along the facial artery, a mean of 4 on each half of the face (range: 2-8), with a mean diameter of 0.94 mm (range: 0.53-1.36 mm) and maximum perforators between 20 and 60 mm from the origin along the length of the facial artery. This roughly corresponds to an area near the angle of the mouth around the nasolabial fold. A local skin flap based on such perforators can be islanded, with greater freedom in flap designing for reconstruction of small-to-moderate-sized intraoral and facial defects in one stage Ethical consideration This study will be approved by the ethics committee of Faculty of Medicine Sohag University. A written informed consent will be taken from every patient that will be included in this study and all patients will be informed about the nature & the aim of the study and the possibility of any complication.

Surgical technique:

After tumor ablation the facial artery perforator along the nasolabial fold was found and marked with a handheld Doppler probe. A perforator near the defect was selected to accomplish a sufficient arc of rotation without tension. The flap was designed to cover the defect based on one perforator and to hide the donor site in the nasolabial fold. An incision on one side of the flap was made to the subcutaneous tissue. Undermining of the flap until the perforators were identified. After the perforators were identified, the flap was redesigned and an incision was made circumferentially. Dissection of the pedicle was performed until tension-free transposition was done to cover the defect, and the distal perforators were sacrificed to help flap movement. For protection against shear forces, the investigators left a small cuff of subcutaneous fat around the perforator

ELIGIBILITY:
Inclusion Criteria:

* Lip defect more than half of lip
* Patients aging 7 to 70 years

Exclusion Criteria:

* Lip defect less than half of lip
* Patients with a major uncontrollable medical illness, chronic heavy smokers

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
change of donor site scar | one year
  the possibility of a one-stage reconstruction and customization. In addition, the use of this flap increases aesthetic results, as it uses a local flap and conceals the donor scar within a natural fold.
  prevent furthur operations for reconstructions. We use( 0..100 visual analog scale) to show change of skin texture to basal line as 0 is the worst result and 100 the best ...patient questionnaire about the result will be done

SECONDARY OUTCOMES:
change of lip size | one year
  as other procedures may cause microstomia and affect speech

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Yossef Elsayed, MD, Study Chair — sohag university , Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ercan A, Ercan LD, Demiroz A. Nasolabial Perforator Flap: A Multi-Tool for Reconstruction of Facial Units. J Craniofac Surg. 2020 Jun;31(4):1042-1045. doi: 10.1097/SCS.0000000000006285. PMID 32168126